CLINICAL TRIAL: NCT04586374
Title: G- Forces On Retrieved ChildrEn Pilot Study
Acronym: G-FORCE
Status: Completed | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 20CS032
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Physiological Shock
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Transported patients with full monitoring (including an arterial line), without inotropic/vasoactive support.
- Study Group: Transported patients with full monitoring and vasoactive/inotropic support being delivered by a syringe driver.

SUMMARY:
G-Forces On Retrieved ChildrEn (Pilot) Study is a feasibility study looking at the effect of G-Forces in vivo during episodes of paediatric critical care transport. The study aims to (i) understand the relationship between the physics of transport on physiological parameters and (ii) assess whether syringe driver delivery (previously demonstrated to be affected by G-forces in vitro), is responsible for physiological variations in transported paediatric patients requiring vasoactive/inotropic infusions.

DETAILED DESCRIPTION:
Throughout the UK, paediatric transport services are responsible for the stabilisation and transport of critically unwell children. This involves moving children from district general hospitals to receive specialist care in tertiary centres and moving children between tertiary and quaternary centres in order to provide the appropriate level of specialist care.

Critically unwell children often require infusions of essential, life-saving medications during episodes of transport. Disruption of these infusions can be destabilising and even life-threatening. Examples of essential infusions include the use of prostin in duct-dependent congenital heart disease, vasoactive/inotropic medications in shock and sedation and muscle relaxants to ensure comfortable, safe transfer.

Critically unwell patients often require support in the form of inotropes/vasopressors to support cardiac contractility and alter vascular tone and are commonly used in the treatment of shock. Physiological response to vasoactive/inotropic drugs is rapid and measurable in terms of cardiovascular status through observing changes in heart rate, blood pressure and oxygenation of peripheral tissues (pulse oximetry). As such these medications offer the potential to observe whether syringe driver delivery variations as mediated through the effect of g-forces exert measurable physiological instability in transported patients.

G-Forces Pilot is a prospective, observational, case-control, feasibility study investigating the effect of G-forces as measured by an accelerometer against physiological parameters of heart rate, invasive blood pressure measurement and oxygen saturations in vivo during episodes of transport. The study aims to understand the relationship between the physics of transport on physiological parameters and to assess whether syringe driver delivery (previously demonstrated to be affected by G-forces in-vitro), is responsible for physiological variations in transported patients requiring vasoactive/inotropic infusions.

The investigators propose to examine this relationship by obtaining and analysing data on physiological parameters in patients during episodes of transport to assess:

(i) Whether G-forces experienced by being in a moving ambulance affect the stability of patient physiological parameters.

(ii) How variations in syringe driver delivery mediated through the effects of G-Forces affect patients in transit as evidenced through instability in physiological parameters whilst receiving vasoactive/inotropic infusions.

This will be examined by the comparison of a control and study group. The control group will consist of patients with full monitoring (including an arterial line), without vasoactive/inotropic support. The study group will consist of patients with full monitoring (including an arterial line) receiving vasoactive/inotropic support through a syringe driver. Data analysis will assess the strength of correlation between patient observations and experienced g-forces recorded during the episode of transport to answer the study question.

ELIGIBILITY:
Inclusion Criteria:

(i) Any child, 36 weeks corrected gestation to 18 years, accepted for transport by the COMET retrieval service who has an arterial line with active arterial blood pressure monitoring at departure from the referring hospital. The decision for the need for an arterial line is determined purely on a clinical basis by the referring, transporting or accepting clinical team.

Exclusion Criteria:

(i) Children outside the specified age range.

(ii) Children who do not have invasive arterial blood pressure monitoring during a transport episode.

(iii) Any case where patients, parents or guardians elect to opt out of data analysis.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Any child, 36 weeks corrected gestation to 18 years, accepted for transport by the COMET retrieval service
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Correlation between physiological parameters and G-forces during transport episode | 12 months study period
  Beat to beat, wave-form data from physiological parameters of heart rate, oxygen saturations and invasive arterial blood pressure measured during transport will provide a set of continuous data outputs. Calculating the correlation coefficient will indicate the strength of relationship between physiological parameters and the experienced G-forces with the aim of answering two questions:
  1. Do G-forces (the acceleration and deceleration forces) experienced by being in a moving ambulance, affect the stability of patient observations - heart rate, blood pressure and oxygen saturations.
  2. Do G-forces experienced by being in a moving ambulance, affect the delivery of vasoactive/inotropic drug infusions which in turn affects the stability of observations.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Shires, BMBS BMedSci, Study Chair — NUH, NHS
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No